CLINICAL TRIAL: NCT00742092
Title: Single Center, Double-blind, Randomized, Placebo-controlled, Two-period/Two-treatment Crossover Study Investigating the Effect of Miglustat on the Nasal Potential Difference in Patients With Cystic Fibrosis Homozygous for the F508del Mutation
Brief Title: Miglustat in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-056A202
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): miglustat
  Interventions: Drug: miglustat
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: miglustat — Oral miglustat capsules 200 mg t.i.d. (three times a day) for 7 days and a single 200 mg dose on Day 8
  Arms: 1
Drug: placebo — Oral placebo capsules matching in appearance miglustat capsules given t.i.d. (three times a day) for 7 days and a single dose on Day 8
  Arms: 2

SUMMARY:
Single Center, Double-Blind, Randomized, Placebo-Controlled, Two-Period/Two-Treatment Crossover Study Investigating the Effect of Miglustat on the Nasal Potential Difference in Patients With Cystic Fibrosis Homozygous for the F508del Mutation

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years and older
* Male or female Non-pregnant women who are to remain non-pregnant for 3 months after the end of the study. Women of childbearing potential must use a reliable method of contraception. Reliable methods of contraception for female patients include the following:
* barrier type devices (e.g., female condom, diaphragm and contraceptive sponge) used ONLY in combination with a spermicide
* intrauterine devices
* oral contraceptive agent
* Depo-Provera™ (medroxyprogesterone acetate)
* levonorgestrel implants Abstention, the rhythm method or contraception by the partner alone are NOT reliable methods of contraception. A woman is considered to have child-bearing potential unless she meets at least one of the following criteria:
* 6 weeks post-surgical bilateral salpingo-oophorectomy or hysterectomy
* Premature ovarian failure confirmed by a specialist gynecologist
* Age > 50 years and not treated with any kind of HRT for at least 2 years prior to screening, and with amenorrhea for at least 24 consecutive months prior to screening and a serum FSH level of > 40 IU/L at screening.
* Age > 55 years and treated with HRT prior to screening with an appropriate medical documentation of spontaneous amenorrhea for at least 24 months. For female patients in the pediatric age range, a reliable method of contraception must be considered, if appropriate.

  * Male patients accepting for the duration of the study and for 3 months thereafter to use a condom and not to procreate a child (not in case of azoospermia)
  * Cystic fibrosis patients homozygous for the F508del mutation as confirmed by genetic test
  * Signed informed consent prior to any study-mandated procedure

Exclusion Criteria:

* Any condition prohibiting the correct measurement of the NPD such as upper respiratory tract infection
* Acute upper respiratory tract or pulmonary exacerbation requiring antibiotic intervention within 2 weeks of screening
* Severe renal impairment (creatinine clearance < 30 mL/min as per Cockroft and Gault)
* Female patients of childbearing potential who will not undergo a pregnancy test prior to enrollment into the study
* History of significant lactose intolerance
* History of neuropathy
* Presence of clinically significant diarrhea (> 3 liquid stools per day for > 7 days) without definable cause within 1 month prior to screening
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease
* FEV1 < 25% of predicted normal
* Oxygen saturation at rest < 88%
* Active or passive smoking as measured using the Smokelyzer®
* Hypersensitivity to miglustat or any excipients
* Planned treatment or treatment with another investigationaldrug or therapy (e.g., gene therapy) within 1 month prior to randomization
* Breast-feeding, pregnant women or women who plan to become pregnant during the course of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The sum of responses in nasal potential difference (NPD) after perfusion with isoproterenol and chloride-free buffer (TCS: Total Chloride Secretion), in the presence of amiloride. | Change from baseline (pre-dose on Day 1) to end-of-treatment (Day 8)

SECONDARY OUTCOMES:
Change in basline nasal potential difference (NPD) response | From baseline (pre-dose on Day 1) to end-of-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lebecque, MD, PhD, Principal Investigator — Catholic University of Louvain
Locations (1):
- Universite Catholique de Louvain, Brussels, Belgium

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834